CLINICAL TRIAL: NCT00158457
Title: Pilot Trial to Evaluate the Efficacy and Tolerance of a Simple Once Daily Combined Regimen Including Tenofovir (TDF), Emtricitabine (FTC) and Efavirenz (EFV) in HIV-1 Infected Patients Naive to Prior Antiretroviral Treatment in Senegal
Brief Title: Simple Once Daily Triple Regimen Including Tenofovir, Emtricitabine and Efavirenz in HIV-1 Infected Patients (ANRS 1207)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Gilead Sciences (Industry); Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 1207; IMEA 025
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-07-03 (Estimated); Status verified 2007-07

CONDITIONS: HIV Infection
Keywords: Simplification regimen; HIV infection; Once a day; Naive patients; Sub-saharian Africa; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Emtricitabine; Racivir; efavirenz

INTERVENTIONS:
Drug: Tenofovir (TDF)
Drug: Emtricitabine (FTC)
Drug: Efavirenz (EFV)

SUMMARY:
In the context of Sub-saharian Africa, this trial evaluate one of the most simple treatment available for HIV-1 infected patients. The combination proposed is a triple antiretroviral therapy with only one intake of 3 pills per day. This combination has already been studied in the North countries.

Here in Senegal, the efficacy and the compliance to treatment will be evaluated after 24, 48 and 96 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Documented infection with HIV-1 (ELISA- Western Blot)
* Outpatient of masculine or feminine gender
* In female patients any risk of pregnancy must be avoid: women at least 1 year past menopause or being confirmed sterile or having an effective contraceptive device
* No previous treatment with antiretroviral therapy
* CDC group C (except tuberculosis if CD4 count is over 350 /ml), CDC group B with CD4+ count under 350/ml and CDC group A with CD4 count under 200/ml.
* Patient has provided informed written consent
* Patient must agree not to take any concomitant medication throughout the duration of the study without first informing the investigator

Exclusion Criteria:

* Deficiency of the patient rendering participation in the study or understanding of the information imparted difficult or even impossible
* Patient participating in a different clinical study
* Presence of serious or developing pathology
* Severe liver failure (TP under 50% et bilirubinemia over 3 LSN)
* Thrombocytopenia with platelet level under 50 000 cells /ml
* Known severe renal pathology (creatinine clearance under 50 ml/min)
* Clinical or biological problem corresponding to indications of grade over or equal 3 of WHO classification
* Karnofsky under 70 percent
* Opportunistic infections
* Patients taking medications not recommended in the context of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-06; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the antiretroviral efficacy as first line treatment assessed as percentage of patients with viral load below 400 copies/ml at week 48 in the intention to treat (ITT) population | S48

SECONDARY OUTCOMES:
Reduction of the viral load and percentage of patients with a viral load lower than 50 copies/ml | S24 and S96
Viral load evolution | S24 and S48
Genotype resistance profile evaluation failing patients | S24, S48, S96
Immune benefits of the combination
Plasma concentrations of FTC, TDF and EFV | S4
Adverse events clinic and lipids
Compliance | S48 and S96

CONTACTS AND LOCATIONS:
Overall Officials: Roland Landman, Study Chair — IMEA- Hôpital Bichat Claude Bernard, France; Papa Salif Sow, Principal Investigator — CHU de Fann, Dakar
Locations (2):
- Senegal (2):
  - Centre de Traitement Ambulatoire, CHU de Fann, Dakar
  - Service des Maladies Infectieuses, CHU de Fann, Dakar